CLINICAL TRIAL: NCT06527586
Title: A Study to Evaluate the Safety and Efficacy of Eye Secret UV Aspheric Silicone Soft (Hydrophilic) 1Day Color Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yung Sheng Optical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUV-01V1.0
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Si-Hy (Otufilcon A) (Experimental)
  Interventions: Device: soft contact lens
- Si-Hy soft contact lens (Active Comparator)
  Interventions: Device: soft contact lens

INTERVENTIONS:
Device: soft contact lens — Vision Correction

SUMMARY:
This was a prospective, randomized, open label, parallel, active-controlled clinical study to assess the safety and efficacy of Silicone Color Contact Lens for vision correction.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 20 to 65.
2. Subject with -1.00 to -10.00 D myopia, less than 1.00 D astigmatism.
3. Subjects must be correctable through spherocylindrical refraction and with soft contact lenses to 0 Log MAR (distance) or better in each eye.
4. Willing to comply with all study procedures and be available for the study duration.
5. Provide signed and dated informed consent form.

Exclusion Criteria:

1. Subjects have a history of allergies that contraindicate contact lens wear.
2. Subjects have other active ocular or systemic diseases such as, but not limited to anterior uveitis (past or present), glaucoma, Sjögren's syndrome, lupus erythematosus, sclerodermas, keratoconus or diabetes.
3. Subjects have medications that would contraindicate contact lens wear.
4. Currently pregnant (to the best of the subject's knowledge), is lactating or is planning a pregnancy within the next 3 months.
5. Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
6. Any active participation in any contact lens or lens care product clinical trial within seven days prior to this study.
7. The presence of clinically significant (grade 3 or 4) anterior segment abnormalities; inflammations such as iritis; or any infection of the eye, lids, or associated structures.
8. Subject has a known history of corneal hypoesthesia (reduced corneal sensitivity), corneal ulcer, corneal infiltrates or fungal infections.
9. Subject has a history of papillary conjunctivitis that has interfered with contact lens wear.
10. Subject has a history of herpetic keratitis retinal detachment or irregular cornea.
11. Subject has a history of recurrent eye or eyelid infections, adverse effects associated with your contact lens wear, intolerance or unusual response to your contact lens wear.
12. The subject has over grade II corneal and conjunctival staining (Oxford scheme) if who has a history of dry eye.
13. Subject had any corneal surgery (e.g., refractive surgery).

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
The effectiveness of corrected visual acuity | 3 Months
  The primary effectiveness endpoint of the study was the comparison of the mean change in logMAR visual acuity (VA) of the subject's worse eye, from baseline (Day 1) to the final visit (3-month), between the groups wearing test lenses and control lenses.

SECONDARY OUTCOMES:
Effectiveness of corrected visual acuity | 1 Week
  The secondary effectiveness endpoint involves comparing the mean difference in LogMAR visual acuity (VA) for each eye-both eyes of each subject-between the test lens and the control lens at one week.

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Linkou-Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No